CLINICAL TRIAL: NCT03329547
Title: An Open-label, Randomised, Single-dose, Two-period Cross-over Study to Evaluate Bioequivalence of SKF101804 Cefixime 400 mg Capsule Versus Cefixime 400 mg Capsule Reference Product in Healthy Adult Participants Under Fasting Conditions
Brief Title: A Bioequivalence Study of SKF101804 Cefixime Versus Cefixime Reference Formulation in Healthy Adults Under Fasting Conditions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in commercial strategy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205732
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Infections, Bacterial
Keywords: Bioequivalence; Pharmacokinetics; SKF101804; Crossover; Cefixime
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: This will be a two-period crossover study. Subjects will receive single oral dose of cefixime 400 mg test capsules and cefixime 400 mg reference capsules in treatment period 1 and 2 under fasting conditions.
Masking Description: This will be an open-label study. Hence, masking will not be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects receiving treatment sequence AB (Experimental): Eligible subjects will receive treatment sequence AB; A= SKF101804 cefixime 400 mg test capsules and B= cefixime 400 mg reference capsules. Subjects will receive single oral dose of treatment A in treatment period 1 on Day 1 and treatment B in treatment period 2 on Day 1. Treatment periods 1 and 2 will be separated by a washout period of 7 to 14 days.
  Interventions: Drug: Cefixime test capsule; Drug: Cefixime reference capsule
- Subjects receiving treatment sequence BA (Experimental): Eligible subjects will receive treatment sequence BA; B= cefixime 400 mg reference capsules and A= SKF101804 cefixime 400 mg test capsules. Treatment periods 1 and 2 will be separated by a washout period of 7 to 14 days. Subjects will receive single oral dose of treatment B in treatment period 1 on Day 1 and A in treatment period 2 on Day 1. Treatment periods 1 and 2 will be separated by a washout period of 7 to 14 days.
  Interventions: Drug: Cefixime test capsule; Drug: Cefixime reference capsule

INTERVENTIONS:
Drug: Cefixime test capsule — SKF101804/cefixime test capsule will be given with a single dose of 400 mg administered orally along with 240 mL of water. It will be available as a dark purple head and off white body locking type capsule with "GSK' printed on cap and "400MG" printed on body of capsule.
Drug: Cefixime reference capsule — Cefixime reference capsule will be given with a single dose of 400 mg administered orally along with 240 mL of water. It will be available as red/orange hard gelatin size 0 capsule with "Cefspan 400 mg" printed on body of capsule.

SUMMARY:
Cefixime is an orally active third generation cephalosporin indicated for the treatment of acute exacerbations of chronic bronchitis, acute otitis media, uncomplicated acute cystitis and uncomplicated pyelonephritis. Cefixime acts by inhibiting the action of proteins involved in the synthesis of bacterial cell walls, which leads to bacterial cell lysis and cell death. Due to lack of bioequivalence between tablet/capsule and suspension formulation of cefixime, consideration needs to be given if the oral suspension is to be substituted for the tablet/capsule. This study is designed to assess whether test SKF101804 cefixime 400 milligrams (mg) capsule is bioequivalent to reference cefixime 400 mg capsule under fasting conditions in healthy adults. Subjects will be randomized in crossover manner to receive single oral doses of treatment A (SKF101804 cefixime test capsules) and treatment B (reference cefixime capsules), followed by a washout period of 7-14 days. Approximately 26 subjects will be included in the study and total duration in the study for each subject will be approximately 5 to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Healthy, non-smoker, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included at investigator discretion in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight within >=50 kilogram (kg) and body mass index (BMI) within the range 19-30 kg per meter square (kg/m^2) (inclusive).
* Healthy male or female subjects. A male subject must agree to use contraception during the treatment period and for at least 5 days after the last dose of study treatment and refrain from donating sperm during this period; a female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Any other condition that is capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal renal function, as determined by creatinine clearance and considered as clinically significant by the investigator will be excluded.
* Abnormal blood pressure as determined by the investigator.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* ALT >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of colitis.
* History of cephalosporin induced hemolytic anemia.
* QT interval corrected for heart rate according to Bazett's formula (QTcB) >450 milliseconds (msec). Subjects with a known risk of QT prolongation will be excluded.
* Past or intended use of over-the-counter or prescription medication including herbal medications, within 14 days prior to dosing unless in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 90 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 90 days before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Presence of Hepatitis B surface antigen (HBsAg) at screening. Positive Hepatitis C antibody test result at screening.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine containing products within 6 months prior to screening.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Known sensitivity to any drugs from the class of cephalosporin, or components thereof.
* Known sensitivity to any drugs from the class of penicillin, or components thereof.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-11 (Estimated); Primary Completion 2018-02-02 (Estimated); Study Completion 2018-02-02 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUC [0-t]) of cefixime test capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime test capsules under fasting conditions.
AUC (0-t) of cefixime reference capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime reference capsules under fasting conditions.
Maximum observed concentration (Cmax) of cefixime test capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime test capsules under fasting conditions.
Cmax of cefixime reference capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime reference capsules under fasting conditions.

SECONDARY OUTCOMES:
AUC from time zero extrapolated to infinite time (AUC [0-infinity]) of cefixime test capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime test capsules under fasting conditions.
AUC(0-infinity) of cefixime reference capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime reference capsules under fasting conditions.
Time of occurrence of Cmax (Tmax) of cefixime test capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime test capsules under fasting conditions.
Tmax of cefixime reference capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime reference capsules under fasting conditions.
Percentage of AUC (0-infinity) obtained by extrapolation (percent AUCex) of cefixime test capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime test capsule under fasting conditions.
Percent AUCex obtained by extrapolation of cefixime reference capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime reference capsules under fasting conditions.
Apparent terminal phase half-life (T1/2) of cefixime test capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime test capsule under fasting conditions.
T1/2 of cefixime reference capsule | Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 20.0 and 24.00 hours post dose
  Blood samples will be collected for pharmacokinetic analysis of cefixime reference capsules under fasting conditions.
Number of subjects with adverse events (AEs) | Up to 27 days
  An AE is any untoward medical occurrence in a clinical study subjects, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Number of subjects with serious AEs (SAEs) | Screening and up to 27 days
  Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Number of subjects with abnormal hematology laboratory parameters as a measure of safety | Up to 27 days
  Hematology parameters will be analyzed including platelet count, red blood cells (RBC) count, hemoglobin and hematocrit level as a measure of safety.
Number of subjects with abnormal biochemistry laboratory parameters as a measure of safety | Up to 27 days
  Biochemistry parameters will be analyzed including blood urea nitrogen (BUN), fasting glucose, potassium, creatinine, sodium, calcium, aspartate aminotransferase (AST)/ serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT), alkaline phosphatase, total and direct bilirubin and total protein as a measure of safety.
Number of subjects with abnormal values for body temperature | Up to 27 days
  Body temperature will be measured in a semi-supine position after at least a 5-min rest.
Number of subjects with abnormal pulse rate | Up to 27 days
  Pulse rate will be measured in a semi-supine position after 5-min rest.
Number of subjects with abnormal respiratory rate | Up to 27 days
  Respiratory rate will be measured in a semi-supine position after at least a 5-min rest.
Number of subjects with abnormal values for blood pressure | Up to 27 days
  Systolic and diastolic blood pressure will be measured in a supine position after 5 minutes rest.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline